CLINICAL TRIAL: NCT06556186
Title: Surgical and Pharmacological Efficacy of Knosp Grade 0-2 Prolactinoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Peking Union Medical College Hospital (Other); West China Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Ningbo Medical Center Lihuili Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0268
Record Dates: First submitted 2024-08-05; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-07

CONDITIONS: Pituitary Tumor
Keywords: pituitary tumor
MeSH Terms: conditions — Pituitary Neoplasms | interventions — Bromocriptine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Operation group (Experimental): Transnasal transsphenoidal pituitary lesion resection under neuroendoscopy
  Interventions: Procedure: Transnasal transsphenoidal pituitary lesion resection under neuroendoscopy
- Drug group (Active Comparator): Bromocriptin 2.5mg, 2-3 times a day
  Interventions: Drug: Bromocriptin 2.5mg, 2-3 times a day

INTERVENTIONS:
Procedure: Transnasal transsphenoidal pituitary lesion resection under neuroendoscopy — Transnasal transsphenoidal pituitary lesion resection under neuroendoscopy
  Arms: Operation group
Drug: Bromocriptin 2.5mg, 2-3 times a day — Bromocriptin 2.5mg, 2-3 times a day
  Arms: Drug group

SUMMARY:
The investigators carried out a multi-center comparative study, involving hospitals including the Second Affiliated Hospital of Zhejiang University School of Medicine, Peking Union Medical College Hospital, West China Hospital, Wenzhou First Hospital, and Li Huili Hospital. This study aimed to compare the efficacy of medication and surgery for specific subtypes of microadenomas and clearly defined macroadenomas (Knosp grades 0-2), in order to determine which is more effective and which has fewer benefits, thereby enhancing the evidence base.

ELIGIBILITY:
Inclusion Criteria:

* Prolactin level greater than three times the normal upper limit
* MRI indicates Knosp Grade 0-2 pituitary adenoma

Exclusion Criteria:

* MRI indicates Knosp grade 3-4 pituitary adenoma
* Taking antidepressants or other psychotropic drugs
* Patients allergic to bromocriptine or cannot tolerate surgery
* Women defined as surgical infertility (i.e. hysterectomy, bilateral salpingectomy, or bilateral oophorectomy), or amenorrhea for more than 2 years
* Critical illness patients, such as those with progressive consciousness disorders, cerebral hernias, and other emergency situations

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
pituitary hormone levels | At 1, 3, 6, 9 and 12 months postoperatively
  Recheck pituitary hormones (PRL, GH, ACTH, etc.)
pituitary MRI | At 1,6 and 12 months postoperatively
  Recheck pituitary MRI

SECONDARY OUTCOMES:
sexual function evaluation | At 1,6 and 12 months postoperatively
  Male:International Index of Erectile Function (IIEF-5); Female:Female Sexual Function Index (FSFI)
menstrual condition | At 6 and 12 months postoperatively
  There is currently no specific "Pituitary Tumor Menstrual Status Questionnaire" for evaluation. The investigators usually evaluate the impact of pituitary tumors on menstruation based on the participants clinical symptoms and the results of sex hormones
lactation | At 1,6 and 12 months postoperatively
  Serum prolactin levels